CLINICAL TRIAL: NCT00365430
Title: SAFE or SORRY? Development and Testing of an Evidence Based Inpatient Safety Program for the Prevention of Common Complications.
Brief Title: SAFE or SORRY? Patient Safety Study of the Prevention of Adverse Patient Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Theo van Achterberg, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SoS245119; 54010002
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Pressure Ulcer; Urinary Tract Infection; Accidental Falls
Keywords: Patient safety; Adverse event; Prevention; Knowledge; Inpatient; Hospital; Nursing home; Long term care; Nurse
MeSH Terms: conditions — Pressure Ulcer; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: safety program — Education, patient involvement, tailored implementation and a computerized registration system

SUMMARY:
The aim of SAFE or SORRY? is to develop and test an evidence based inpatient safety program for the prevention of three frequently occuring adverse events: pressure ulcers, urinary tract infections and falls.

DETAILED DESCRIPTION:
Background Patients in hospitals and nursing homes are at risk for the development of, often preventable, somatic complications. However, preventive care is not always optimal. Although guidelines are available for many complications, compliance with the guidelines appears to be lacking. Besides general barriers that inhibit implementation, this non-compliance is also associated with the large number of guidelines competing for attention. As implementation of a guideline is time-consuming, organisations can never implement all available guidelines. Another problem is lack of feedback about performance using clear quality indicators and lack of a recognizable, unambiguous system for implementation.

Aim The aim of SAFE or SORRY? is to develop and test an evidence based inpatient safety program for the prevention of three frequently occuring adverse events: pressure ulcers, urinary tract infections and falls.

Participants Patients and nurses will be recruited from ten hospital wards and ten nursing home wards in the Netherlands. All nurses and all adult patients who are admitted for more than three days, will be asked for informed consent.

Method This study consists of two phases. In the first phase the program will be developed. The content of the program is based on the evidence based guidelines on pressure ulcers, urinary tract infections and falls. The program consists of a computerized registration and feedback system, an educational program for nurses and caregivers, and educational material for the patients.

In the second phase the program will be tested in a cluster randomised clinical trial. The program will be implemented on ten wards (5 hospital wards and 5 nursing home wards), i.e. the intervention group. The control group will continue to give care as usual.

Outcome measures Primary outcome measure: incidence of pressure ulcers, urinary tract infections and falls Secondary outcome measures: Utilization of preventive interventions and knowledge of nurses and caregivers regarding the complications and their prevention.

ELIGIBILITY:
Inclusion Criteria:

* patients on participating wards admitted for more than three days
* all nurses on participating wards

Exclusion Criteria:

* students on participating wards

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (count incidence of Pressure Ulcers, Urinary Tract Infections, and Falls | nine months

SECONDARY OUTCOMES:
Utilization of preventive interventions and knowledge of nurses and caregivers | nine months

CONTACTS AND LOCATIONS:
Overall Officials: Theo van Achterberg, PhD, Study Director — Scientific Institute for Quality of Healthcare (IQ Healthcare), Radboud University Nijmegen Medical Center
Locations (10):
- Netherlands (10):
  - Alysis Zorggroep lokatie Rijnstate, Arnhem, Gelderland
  - Zorggroep Maas en Waal, Beneden-Leeuwen, Gelderland
  - Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Radboud University Nijmegen Medical Center, Nijmegen, Gelderland
  - Stichting De Waalboog, Nijmegen, Gelderland
  - Zorggroep Zuid-Gelderland, Nijmegen, Gelderland
  - Universitair Longcentrum Dekkerswald, Nijmegen, Gelderland
  - Zorggroep Noord-Limburg Venlo, Venlo, Noord-Limburg
  - Stichting SVVE De Archipel, Eindhoven, North Brabant
  - Stichting De Riethorst Stromenland, Geertruidenberg, North Brabant

REFERENCES:
- [Derived] van Gaal BG, Schoonhoven L, Mintjes JA, Borm GF, Hulscher ME, Defloor T, Habets H, Voss A, Vloet LC, Koopmans RT, van Achterberg T. Fewer adverse events as a result of the SAFE or SORRY? programme in hospitals and nursing homes. part i: primary outcome of a cluster randomised trial. Int J Nurs Stud. 2011 Sep;48(9):1040-8. doi: 10.1016/j.ijnurstu.2011.02.017. Epub 2011 Mar 17. PMID 21419411
- [Derived] van Gaal BG, Schoonhoven L, Vloet LC, Mintjes JA, Borm GF, Koopmans RT, van Achterberg T. The effect of the SAFE or SORRY? programme on patient safety knowledge of nurses in hospitals and nursing homes: a cluster randomised trial. Int J Nurs Stud. 2010 Sep;47(9):1117-25. doi: 10.1016/j.ijnurstu.2010.02.001. Epub 2010 Mar 3. PMID 20202633
- [Derived] van Gaal BG, Schoonhoven L, Hulscher ME, Mintjes JA, Borm GF, Koopmans RT, van Achterberg T. The design of the SAFE or SORRY? study: a cluster randomised trial on the development and testing of an evidence based inpatient safety program for the prevention of adverse events. BMC Health Serv Res. 2009 Apr 1;9:58. doi: 10.1186/1472-6963-9-58. PMID 19338655
- See also: Guideline prevention urinary tract infection (The Netherlands) — http://www.wip.nl/free_content/richtlijnen/11111111blaaskatheterisatie.pdf
- See also: Guideline Urinary Tracts Infections (The Netherlands) — http://www.verpleeghuisartsen.nl